CLINICAL TRIAL: NCT06094075
Title: Effectiveness of an Individualized Training Based on Dynamic Strength Index on Sprinting, Jumping and Change of Direction Performance in Basketball Players: a Randomized Controlled Trial.
Brief Title: Dynamic Strength Index-based Intervention in Basketball.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: Middlesex University (Other)
Responsible Party: Principal Investigator, Žiga Kozinc, Assistant professor and research fellow, University of Primorska
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DSI_Intervention_FVZ
Record Dates: First submitted 2023-10-12; First posted 2023-10-23 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Sports; Basketball; Strength Training

STUDY DESIGN:
Intervention Model Description: Two groups (randomization used for allocation), tested before and after the intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSI-based training group (Experimental): This group will perform resistance exercises based in their DSI values.
  Interventions: Other: Resistance training based on DSI value
- Normal training group (Active Comparator): This group will perform a normal, typical resistance exercise program
  Interventions: Other: Normal training group

INTERVENTIONS:
Other: Resistance training based on DSI value — The intervention consist of modifying the ongoing resistance exercises. Those with low DSI values will perform ballistics, explosive exercises. Those with high DSI will perform heavy-load training. The resistance training program will consist of 2 sessions per week for 5 weeks (10 sessions in total). The sessions will be separated by a minimum of 48 hours. The strength training group will consist mostly of exercises with high load, whereas the ballistic training group will perform ballistic exercises with low load or without any additional load. The training principle will be the same for both subgroups, consisting of 3 exercises per training session and a total of 6 exercises per week, with four of the exercises being bilateral, one unilateral, and one quasi-unilateral (Bulgarian split squat and scissor jumps).
  Arms: DSI-based training group
Other: Normal training group — The participants will do a general training program (not based on DSI values). The resistance training program will consist of 2 sessions per week for 5 weeks (10 sessions in total). The sessions will be separated by a minimum of 48 hours. The strength training group will consist mostly of exercises with high load, whereas the ballistic training group will perform ballistic exercises with low load or without any additional load. The training principle will be the same for both subgroups, consisting of 3 exercises per training session and a total of 6 exercises per week, with four of the exercises being bilateral, one unilateral, and one quasi-unilateral (Bulgarian split squat and scissor jumps).
  Arms: Normal training group

SUMMARY:
The goal of this randomized controlled trial will be to determine the effectiveness of the dynamic strength index (DSI) in optimizing training programs to improve physical performance proxies (sprinting, jumping, and CoD) in basketball players. Subjects will be randomly allocated to one of two groups: the intervention group and the control group. Measurement and intervention will occur during a 7-week in-season period, right before the play off starts. Throughout this period, all participants will engage in an average of 10 hours of basketball training per week, which will comprise 5 basketball sessions and 2 strength training sessions. In addition, they are anticipated to play 2 games weekly. A pre-test will be performed one week before the first training session, and post-tests will be performed in the week after the training sessions have finished. Athletes will perform both testing sessions at the same time of the day (± 2 hours). Each athlete will perform a 20-m sprint test, with timing gates positioned at every 5 m distance, a 505 CoD test, countermovement jump (CMJ), and isometric mid-thigh pull (IMTP). Based on CMJ peak force and IMTP peak force data, we will calculate DSI. Based on the average DSI value, the participants in the intervention group will be divided into two groups - strength group and ballistic group.

ELIGIBILITY:
Inclusion Criteria:

* Perform basketball training for at least 5 years
* Plays in professional regional, national or international league

Exclusion Criteria:

* Any musculoskeletal injury in the past 6 months
* Any neurological issues
* Any chronic non-communicable diseases

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
20 m Sprint performance | Baseline and after 5 weeks.
  20 m sprint test in seconds
Change of direction performance | Baseline and after 5 weeks.
  Standardized 505-agility test
Jumping ability | Baseline and after 5 weeks.
  Jump height during jumps with countermovement

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided